CLINICAL TRIAL: NCT00864435
Title: A Two-Way Crossover, Open-Label, Single Dose, Fasting, Bioequivalence Study of Carvedilol 12.5 mg Tablets Versus Coreg® 12.5 mg Tablets in Normal, Healthy, Non-Smoking Male and Female Subjects
Brief Title: A Relative Bioavailability Study of Carvedilol 12.5 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 3159
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Carvedilol; Healthy subjects
MeSH Terms: interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Carvedilol 12.5 mg Tablets, single dose
  Interventions: Drug: Carvedilol 12.5 mg Tablets, single dose
- B (Active Comparator): Coreg® 12.5 mg Tablets , single dose
  Interventions: Drug: Coreg® 12.5 mg Tablets , single dose

INTERVENTIONS:
Drug: Carvedilol 12.5 mg Tablets, single dose — A: Experimental Subjects received Shasun Chemicals and Drugs Ltd. formulated products under fasting conditions
  Arms: A
Drug: Coreg® 12.5 mg Tablets , single dose — B: Active comparator Subjects received GlaxoSmithKline, USA formulated products under fasting conditions
  Other Names: Carvedilol
  Arms: B

SUMMARY:
To compare the rate and extent of absorption of carvedilol from a test formulation of Carvedilol 12.5 mg Tablets versus the reference Coreg® 12.5 mg Tablets under fasting conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Two-way crossover, randomized, open-label, single-dose, fasting, bioequivalence study

Official Title: A Two-Way Crossover, Open-Label, Single Dose, Fasting, Bioequivalence Study of Carvedilol 12.5 mg Tablets Versus Coreg® 12.5 mg Tablets in Normal, Healthy, Non-Smoking Male and Female Subjects

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking male or female with a minimum age of 18 years.
2. Body Mass Index (BMI = weight/heigh2) greater than or equal to 18.5 kg/m2 and less than or equal to 29.9 kg/m2
3. Normal findings in the physical examination, 12-lead ECG and vital signs (blood pressure between 106-140/66-90 mmHg, heart rate between 60-99 beats/minute, temperature between 35.8°C and 37.5°C)
4. Negative for drugs of abuse and nicotine.
5. Negative for hepatitis B-surface antigen, hepatitis C and HIV.
6. Female subjects: negative for pregnancy (as evaluated by serum ß-CG test).
7. No clinical laboratory values outside of the acceptable range as defined by BCR, unless the Principal Investigator decides that they are not clinically significant.
8. Female subjects who were surgically sterile for at least 6 months or post-menopausal for at least 1 year, or avoided pregnancy for at least 10 days before the study, during the study and up until 1 month after the end of the study.
9. Availability of the subject for the entire study period and willingness of the subject to adhere to protocol requirements, as evidenced by a signed ICF

Exclusion Criteria:

1. Known history of hypersensitivity to carvedilol (e.g. Coreg®) and/or related beta¬blockers such as propranolol (Inderal®, nadolol (Corgard®), labetalol (Trandate®, metoprolol (Lopressor®, Betaloc®, atenolol (Tenormin®, sotalol, timolol, pindolol, or acebutolol.
2. Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, hematological, liver or kidney disease, unless deemed not clinically significant by the Principal Investigator or Sub-investigator.
3. Presence of any significant physical or organ abnormality.
4. Any history or evidence of psychiatric or psychological disease (including depression) unless deemed not clinically significant by the Principal Investigator or Sub-investigator.
5. Known history of frequent headaches or migraines.
6. Known history of chronic bronchitis or any bronchospastic condition.
7. Any clinically significant illness during the 4 weeks before this study.
8. Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
9. Any history of severe allergic reaction (including drugs, food, insect bites, environmental allergens).
10. Significant or recent history of asthma (after 12 years of age).
11. Any subject with a history of drug abuse.
12. Any subject with a recent (less than 1 year) history of alcohol abuse.
13. Use of any prescription medication within 14 days preceding this study.
14. Use of any over-the-counter (OTC) cough and cold medication containing dextromethorphan within 14 days preceding this study.
15. Use of OTC medication within 7 days preceding this study (except for spermicidal/barrier contraceptive products).
16. Female subjects: use of contraceptives (oral, emergency [plan B®, transdermal, implant, Mirena® IUD, NuvaRing®) within 30 days before drug administration or a depot injection of progestogen drug (e.g. Depo-Provera® within 1 year before drug administration.
17. Female subjects: evidence of pregnancy or lactation.
18. Any subject who had blood drawn within 56 days preceding this study, during the conduct of any clinical study at a facility other than BCR, or within the lockout period specified by a previous study conducted at BCR.
19. Participated in a clinical trial with an investigational drug within 30 days preceding this study.
20. Any subject who had donated blood within 56 days preceding this study.
21. Any subject who had participated as a plasma donor in a plasmapheresis program within 7 days preceding this study.
22. Intolerance to venipuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Y. Tam,, MD, Principal Investigator — Biovail Contract Research
Locations (1):
- Biovail Contract Research (A Division of Biovail Corporation), Toronto, Ontario, Canada